CLINICAL TRIAL: NCT06661096
Title: Temporomandibular Joint Dysfunction (TMJD)
Brief Title: Comparative Study Between Level I and Level II Temporomandibular Joint Arthroscopy in Wilkes Stage III Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Gamal Thabet (Other)
Responsible Party: Sponsor-Investigator, Mohamed Gamal Thabet, principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMJ arthroscopy
Record Dates: First submitted 2024-10-21; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMJ dysfunction (Experimental): TMJ arthroscopy
  Interventions: Procedure: TMJ arthroscopy

INTERVENTIONS:
Procedure: TMJ arthroscopy — level I and level II TMJ arthroscopy

SUMMARY:
Temporomandibular joint dysfunction (TMJD) represents a common health problem. Its prevalence is nearly 31% in adults and 11% in adolescence, more common in females. Aetiologies of TMJD are multifactorial and can be attributed to both physical and psycho-social factors. Internal derangement of the temporomandibular joint (TMJ) is the most frequent disorder; with anterior disc displacement is the most common form. Wilkes has classified internal derangement into five stages; patients with stage III usually present with limited mouth opening, joint pain and deviation of jaw upon opening to the affected side. MRI is considered the gold standard for diagnosis. Treatment of TMJD include non-surgical and surgical methods. Non-surgical treatment includes instructions, pharmacotherapy, physiotherapy and occlusal splints; while surgical interventions include minimally invasive procedures (arthroscopy and arthrocentesis) and open joint surgery

DETAILED DESCRIPTION:
Arthroscopy of TMJ was first introduced by Ohnishi in 1975. There are three different levels of TMJ arthroscopy. Level I, single puncture arthroscopy, it allows lysis of adhesions in the upper joint compartment and lavage of the joint space and the inflammatory products. Level II is done by double puncture and it enables to perform maneuvers such as lateral pterygoid myotomy and ablation of the retrodiscal tissue. Operative devices including arthroscopic instruments, Nd-YAG and Holmium laser, and the high-frequency wave system (Coblation) is very useful for tissue coagulation and cutting. Both levels enabled getting joint mobilization and significant pain reduction. Level III (arthroscopic discopexy), it needs customized special instruments.

ELIGIBILITY:
Inclusion Criteria:

* Wilkes stage III patients

Exclusion Criteria:

* previous TMJ surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-13 (Actual); Primary Completion 2025-10-13 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
maximum inter-incisal opening | 6 months
  change of maximum inter-incisal opening, in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gamal Thabet, MD, Principal Investigator — MGThabet
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No